CLINICAL TRIAL: NCT07105553
Title: Neuro Glove: A Prospective Self-Controlled Study of Glove Compression as a Protective Strategy Against Chemotherapy-Induced Peripheral Neuropathy in Women With Gynecologic Malignancies
Brief Title: Glove Compression for Chemotherapy-Induced Neuropathy
Acronym: NEURO-GLOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Principal Investigator, Ankara Etlik City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AEŞH-EK1-2023-828; AEŞH-EK1-2023-828 (Registry Identifier: Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-07-13; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN); Gynecologic Cancers; Ovarian Cancer (OvCa); Endometrial Cancer
Keywords: Peripheral Neuropathy; CIPN; Taxane Toxicity; Surgical Glove Compression; Supportive Care in Oncology; EORTC QLQ-CIPN20; Gynecologic Malignancy
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention, consisting of tight-fitting surgical gloves worn on the non-dominant hand during paclitaxel infusion. The dominant hand serves as an internal control for each participant. This single-group, self-controlled design allows intra-individual comparison of neuropathy outcomes.
Masking Description: This is an open-label study; no parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Cohort - Self-Controlled (Experimental): This arm includes female patients with gynecologic malignancies receiving paclitaxel-based chemotherapy. Each participant's non-dominant hand received the intervention of two tight-fitting surgical gloves (one size smaller than standard), while the dominant hand remained ungloved and served as an internal control. The gloves were worn during each paclitaxel infusion, starting 30 minutes before the infusion and removed 30 minutes after completion. Neuropathy was assessed using the EORTC QLQ-CIPN20 questionnaire at baseline, after cycle 3, and at the end of treatment. No additional clinical visits were scheduled outside of routine oncology care.
  Interventions: Device: Surgical Glove Compression

INTERVENTIONS:
Device: Surgical Glove Compression — Participants wore two tight-fitting surgical gloves (one size smaller than standard) on the non-dominant hand. The gloves were applied 30 minutes prior to each paclitaxel infusion, remained in place during the infusion, and were removed 30 minutes afterward. The dominant hand remained ungloved and served as an internal control. This intervention was entirely non-pharmacologic and was integrated into routine chemotherapy sessions.
  Other Names: Physical Compression Using Tight-Fitting Gloves

SUMMARY:
This study investigates whether wearing tight-fitting surgical gloves on the non-dominant hand could help prevent chemotherapy-induced peripheral neuropathy (CIPN) in women with gynecologic cancers treated with paclitaxel. In this prospective, self-controlled observational study, seventy-six patients wear two tight surgical gloves on their non-dominant hand during each paclitaxel infusion. The dominant hand, without gloves, serves as a control. Neuropathy symptoms are assessed using the EORTC QLQ-CIPN20 questionnaire at baseline, mid-treatment, and end of treatment. Electromyography (EMG) is performed if clinically indicated.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common, dose-limiting, and often persistent adverse effect of taxane-based chemotherapy, particularly in women with gynecologic malignancies. CIPN significantly impairs quality of life and may necessitate chemotherapy dose reductions or discontinuation. Despite its clinical relevance, no pharmacologic agent has been proven to prevent CIPN. Accordingly, non-pharmacologic strategies such as physical compression have gained attention as potential neuroprotective interventions.

This prospective, non-randomized, self-controlled observational study is being conducted at Etlik City Hospital, Ankara, Türkiye. A total of seventy-six female patients aged 18 years or older with histologically confirmed gynecologic cancers (endometrial and ovarian) scheduled to receive six cycles of carboplatin-paclitaxel chemotherapy was enrolled. The intervention involves applying two tight-fitting surgical gloves (one size smaller than standard) to the non-dominant hand starting 30 minutes before each paclitaxel infusion, worn throughout the infusion, and removed 30 minutes afterward. The dominant hand, without compression, serves as an internal control.

Peripheral neuropathy symptoms are assessed using the EORTC QLQ-CIPN20 questionnaire, a validated tool developed by the European Organisation for Research and Treatment of Cancer. The Turkish version has been previously validated. The CIPN20 includes twenty items scored on a 1 (not at all) to 4 (very much) Likert scale, yielding a total score range from 20 to 80. CIPN20 assessments are conducted at baseline (prior to treatment), after cycle three, and after cycle six. Neurological consultation and electromyography (EMG) are performed only in patients reporting significant neuropathic symptoms and if clinically indicated.

All data collection occurs during routine clinical visits. The study remains entirely non-interventional and is integrated into standard oncology care without additional diagnostic or procedural burdens to participants. The primary objective is to evaluate the feasibility and potential role of glove compression in mitigating CIPN development in the intervention hand compared to the control hand, using validated patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years
* Histologically confirmed gynecologic malignancy (e.g., ovarian, or endometrial cancer)
* Scheduled to receive carboplatin-paclitaxel chemotherapy administered every 21 days
* Planned for a total of six chemotherapy cycles
* ECOG performance status 0-2
* Ability to provide written informed consent

Exclusion Criteria:

* Patients receiving neoadjuvant chemotherapy with planned surgery
* Patients receiving weekly (dose-dense) paclitaxel regimens
* Prior exposure to neurotoxic chemotherapy agents (e.g., taxanes, platinum compounds, proteasome inhibitors, anti-tubulin agents)
* History of pre-existing peripheral neuropathy
* Known allergy to latex or surgical gloves
* Diagnosed peripheral vascular disease
* Concurrent use of medications that may mask or modulate neuropathy symptoms (e.g., gabapentinoids, SNRIs, vitamin B complex, alpha-lipoic acid)
* Clinical diagnosis of diabetic neuropathy or history of alcohol-related neuropathy
* Raynaud's phenomenon or other cold-sensitive vascular conditions
* Other neurological disorders that may interfere with neuropathy assessment
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade ≥2 Chemotherapy-Induced Peripheral Neuropathy (CIPN) in the Intervention vs. Control Hand | At Day 1 (baseline, prior to chemotherapy), Day 64 (after Cycle 3), and Day 127 (after Cycle 6); each chemotherapy cycle is 21 days.
  Peripheral neuropathy severity will be assessed using the validated EORTC QLQ-CIPN20 questionnaire. The sensory subscale score ranges from 0 to 100, with higher scores indicating worse symptoms. A total score of ≥25 will be defined as grade 2 or higher neuropathy. Each patient will serve as their own control: the non-dominant hand will receive the surgical glove compression intervention, while the dominant hand will not. The difference in incidence of grade ≥2 neuropathy between the two hands will be evaluated.
  Unit of Measure: Percentage of patients with grade ≥2 neuropathy, defined as a sensory score ≥25 on the EORTC QLQ-CIPN20 (range 0-100; higher scores indicate worse symptoms).

SECONDARY OUTCOMES:
Incidence of Grade ≥2 Chemotherapy-Induced Peripheral Neuropathy by Baseline Weight Loss Status | From baseline (Day 1) to end of treatment (Day 127, after Cycle 6); each cycle is 21 days.
  Peripheral neuropathy severity will be assessed using the validated EORTC QLQ-CIPN20 questionnaire. Scores range from 0 to 100, with higher scores indicating worse symptoms. A total sensory score ≥25 will be defined as grade 2 or higher neuropathy. This outcome evaluates whether baseline weight loss of ≥10% is associated with the development of grade ≥2 CIPN at the end of treatment. Analyses will include multivariate regression models.
  Unit of Measure: Percentage of patients with grade ≥2 CIPN (EORTC QLQ-CIPN20 score ≥25)
Incidence of Grade ≥2 Chemotherapy-Induced Peripheral Neuropathy by ECOG Performance Status | From baseline (Day 1) to end of treatment (Day 127, after Cycle 6); each cycle is 21 days.
  Peripheral neuropathy severity will be assessed using the validated EORTC QLQ-CIPN20 questionnaire. Scores range from 0 to 100, with higher scores indicating worse symptoms. A total sensory score ≥25 will be defined as grade 2 or higher neuropathy. This outcome evaluates whether ECOG performance status is associated with the development of grade ≥2 CIPN at the end of treatment. Analyses will include multivariate regression models.
  Unit of Measure: Percentage of patients with grade ≥2 CIPN (EORTC QLQ-CIPN20 score ≥25)
Change in EORTC QLQ-CIPN20 Sensory Score Over Time | At Day 1 (baseline, prior to chemotherapy), Day 64 (after Cycle 3), and Day 127 (after Cycle 6); each chemotherapy cycle is 21 days.
  Peripheral neuropathy will be assessed using the validated EORTC QLQ-CIPN20 sensory subscale, which ranges from 0 to 100, with higher scores indicating worse symptoms. This outcome measures the change in sensory score from baseline to mid-treatment (Week 9) and post-treatment (Week 18), comparing the intervention (gloved) and control (non-gloved) hands.
  Unit of Measure: Mean change in sensory score (range 0-one hundred)
Change in Quality of Life Based on EORTC QLQ-C30 Global Health Status | From baseline (Day 1) to end of treatment (Day 127, after Cycle 6); each cycle is 21 days.
  Quality of life will be assessed using the Global Health Status subscale of the validated EORTC QLQ-C30 questionnaire. Scores range from 0 to 100, with higher scores indicating better quality of life. This outcome measures the change in Global Health Status scores from baseline to the end of treatment.
  Unit of Measure: Mean change in Global Health Status score (range 0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No